CLINICAL TRIAL: NCT06819319
Title: A Phase II Study of SHR-A2102 in Combination With Adebrelimab as Neoadjuvant Therapy for Early Triple-Negative Breast Cancer
Brief Title: SHR-A2102 Combined With Adebrelimab as Neoadjuvant Therapy for Early Triple-Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-023; BC-NEO-IIT-SHR-A2102-SHR1316 (Other: Protocol Number)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Treatment group (Experimental): Subjects will receive four cycles of SHR-A2102 combined with adebrelimab therapy. Before the fifth cycle, efficacy is evaluated. If the response is PR/CR, the original regimen will be continued for another four cycles. If SD/PD or PR but deemed unbeneficial by the investigator, treatment will be switched to four cycles of TCb combined with pembrolizumab.
  Interventions: Drug: SHR-A2102 ; Adebrelimab injection

INTERVENTIONS:
Drug: SHR-A2102 ; Adebrelimab injection — SHR-A2102 is administered intravenously, Adebrelimab is administered intravenously

SUMMARY:
This is a prospective, open-label, multicenter Phase II study evaluating the efficacy and safety of of SHR-A2102 in combination with Adebrelimab in Early Triple-Negative Breast Cancer(TNBC)

DETAILED DESCRIPTION:
This study plans to enroll patients with early-stage TNBC. The patients will first receive 8 cycles of neoadjuvant therapy, with imaging examinations conducted every 2 cycles to evaluate the treatment response. Subjects who complete the 8 cycles and are suitable for surgery will undergo surgical treatment after the completion of neoadjuvant therapy. The postoperative adjuvant therapy will last for one year. Subjects will continue medication until surgery is completed, or until disease progression, intolerable toxicity, withdrawal of informed consent, or when the investigator determines that medication must be terminated.

ELIGIBILITY:
3.1 Inclusion Criteria

Subjects must meet all of the following criteria to be eligible:

Age and gender: Female, ≥18 years old.

Histopathological confirmation:

Invasive breast cancer confirmed by histopathology.

No prior systemic anti-tumor therapy for breast cancer.

Triple-negative PD-L1-positive breast cancer:

ER/PR-negative (IHC nuclear staining <10%).

HER2-negative (IHC 0/1+ without FISH testing or IHC 2+ with FISH-negative amplification).

PD-L1 Combined Positive Score (CPS) ≥1.

Tumor stage: T1c-T2, N0-1 or T1a-T1b, N1 (per AJCC 8th Edition criteria).

Measurable lesion: At least one measurable target lesion per RECIST v1.1.

ECOG performance status: 0-1.

Life expectancy: ≥3 months.

Adequate organ and bone marrow function (within 1 month prior to treatment, without corrective therapy within 14 days before first dose):

Bone marrow:

Absolute neutrophil count (ANC) ≥2.0 ×10^9/L.

Platelets ≥100 ×10^9/L.

Hemoglobin ≥100 g/L.

Liver/kidney function:

Albumin ≥3.0 g/dL.

Total bilirubin <1.5 × ULN.

ALT/AST <1.5 × ULN.

Alkaline phosphatase ≤2.5 × ULN.

BUN and serum creatinine <1.5 × ULN or creatinine clearance >60 mL/min (Cockcroft-Gault formula).

Coagulation: PT and APTT ≤1.5 × ULN.

Cardiac function: LVEF ≥55% by echocardiography (ECHO).

QT interval: QTcF ≤470 ms.

Reproductive status:

Premenopausal women: Negative serum pregnancy test within 14 days before treatment.

Non-lactating.

All subjects must use effective barrier contraception during treatment and for 6 months post-treatment.

Informed consent: Willing to sign informed consent and comply with study procedures.

3.2 Exclusion Criteria

Subjects meeting any of the following criteria will be excluded:

Unconfirmed diagnosis: Breast cancer not histopathologically confirmed.

Specific subtypes: Bilateral, inflammatory, or occult breast cancer.

Metastatic disease: Evidence of metastatic breast cancer (excluded via chest/abdominal CT and bone scan; PET/CT allowed as alternative).

Prior anti-tumor therapy:

Chemotherapy, radiotherapy, targeted therapy, or endocrine therapy for breast cancer.

Curative radiotherapy within 4 weeks or palliative radiotherapy within 2 weeks before first dose.

Prior immunotherapy: Anti-PD-1, anti-PD-L1, anti-PD-L2, or other immune checkpoint inhibitors.

Concurrent anti-tumor therapy: Any other anti-cancer treatments during the study.

Second primary malignancy: Except adequately treated non-melanoma skin cancer.

Transplant history: Prior organ or bone marrow transplantation.

Recent clinical trials: Participation in another drug trial within 4 weeks prior to enrollment.

Immunosuppressive therapy: Systemic corticosteroids (>10 mg/day prednisone equivalent) or immunosuppressants within 2 weeks before first dose (excluding inhaled/topical steroids).

Vaccination: Live or attenuated vaccines within 4 weeks before first dose.

Major surgery: Non-breast-related major surgery within 4 weeks before first dose or incomplete recovery.

Autoimmune diseases:

Active autoimmune disease or history of autoimmune disease with potential recurrence (e.g., autoimmune hepatitis, uveitis, thyroid dysfunction requiring systemic treatment).

Exceptions: Vitiligo, psoriasis, alopecia, controlled childhood asthma, or type 1 diabetes managed with insulin.

Immunodeficiency: HIV-positive, congenital/acquired immunodeficiency disorders.

Cardiovascular disease:

History within 6 months: Myocardial infarction, stroke (excluding lacunar infarct), pulmonary embolism, unstable angina, NYHA Class III/IV heart failure.

Clinically significant arrhythmia, primary cardiomyopathy, atrial fibrillation (EHRA ≥2b), uncontrolled hypertension, or QTcF >470 ms.

Pulmonary disease:

Interstitial lung disease, idiopathic pulmonary fibrosis, severe COPD/asthma, or autoimmune/collagen vascular diseases with pulmonary involvement.

Infections:

Active hepatitis B (HBsAg+ with HBV DNA ≥500 IU/mL), hepatitis C (HCV RNA > ULN), cirrhosis, or severe infections requiring antimicrobial therapy.

Bleeding/thrombosis disorders: Hereditary/acquired bleeding or thrombotic tendencies (e.g., hemophilia).

Hypersensitivity: Allergy or contraindication to study drug components.

Pregnancy/lactation: Pregnant, breastfeeding, or unwilling to use contraception.

Comorbidities: Uncontrolled conditions (e.g., hypertension, diabetes, active infections) contraindicating ADC or PD-L1 inhibitors.

Neurological/psychiatric disorders: Epilepsy, dementia, or other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
PCR rate | At the time of surgery
  Total pathological complete response (tpCR: ypT0-is，ypN0)

SECONDARY OUTCOMES:
EFS | 3-10 years
  Event-free survival (EFS)
DFS | 5-10 years
  Disease-free survival (DFS)
DDFS | 5-10 years
  Distant disease-Free Survival (DDFS)